CLINICAL TRIAL: NCT06904885
Title: Implementing a Guideline-based Model of Care for Hip and Knee Osteoarthritis in Finland. A Benchmarking-controlled Trial (FIN-OA)
Acronym: FIN-OA
Status: Not yet recruiting | Type: Observational
Sponsor: University of Jyvaskyla (Other)
Collaborators: University of Southern Denmark (Other); University of Oulu (Other); University of Helsinki (Other); Tampere University (Other); University of Limerick (Other)
Responsible Party: Principal Investigator, Riikka Holopainen, Visiting researcher, University of Jyvaskyla
Other Study IDs: 263/13.00.04.00/2025
Record Dates: First submitted 2025-03-03; First posted 2025-04-01 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis of the Hip or Knee
Keywords: osteoarthritis; implementation; benchmarking controlled trial; model of care; care pathway
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis | interventions — Papaverine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Patients participating GLA:D program
- GLA:D -trained physiotherapists
  Interventions: Behavioral: Implementation of a guideline-based model of care for hip and knee osteoarthritis
- Registry data from national registries (pre): Data of people with hip or knee OA from national registries from all Wellbeing Services Counties in Finland before the implementation of new model of care.
- Registry data from national registries (post): Data of people with hip or knee OA from national registries from all Wellbeing Services Counties in Finland after the implementation of new model of care.

INTERVENTIONS:
Behavioral: Implementation of a guideline-based model of care for hip and knee osteoarthritis — Guideline-based model of care including GLA:D (Good Life with osteoArthritis from Denmark) -program that includes training for physiotherapists and group based education and exercise for patients with hip and knee OA.
  Groups: GLA:D -trained physiotherapists

SUMMARY:
This project aims to bridge the gap between guideline recommendations and clinical practice in osteoarthritis (OA) management. By implementing a systematic, evidence-based model of care, the project seeks to improve patient outcomes, reduce healthcare costs, and provide equitable access to care. The project consists of three phases. In the first phase the current OA care is mapped through registry review and questionnaires and interviews of patients and healthcare professionals. In the second, implementation phase of the project, a plan will be created how to support healthcare professionals in delivering care according to the new model of care and training and support will be offered according to the plan. In the third phase of the project, the implementation success will be evaluated, and the costs of OA care evaluated and compared to baseline data. In addition, patient-reported data will be collected from those patients, who participate in the group-based exercise and education program.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a growing global health challenge, due to the significant increase in prevalence of knee and hip OA. In Finland, OA care costs are substantial, driven by diagnostic procedures, medical treatments, and indirect costs such as work absenteeism. The international guidelines recommend education, exercise, and weight management as first-line treatment options, but adherence to guidelines is inconsistent. This project aims to explore regional differences in OA care and beliefs and OA care practices in Finland. In addition, we will implement and evaluate a guideline-based model of care for hip and knee OA, that includes the Good Life with osteoarthritis from Denmark (GLA:D®) program as the preferred non-surgical management option in local care pathways. In addition, the aim is to share evidence-based OA knowledge and management skills nationwide.

This study is a hybrid type-3 benchmarking-controlled implementation trial. It is nested in primary healthcare in two Wellbeing Services Counties. The study includes three phases: pre-implementation, implementation, and evaluation. The pre-implementation activities include mapping the current OA care through registry review (healthcare utilization and costs from 2019-2024). In addition questionnaires and interviews of patients and healthcare professionals (beliefs and practices) will be conducted. Planned activities of the implementation phase include developing and integrating a new model of care (including GLA:D®) into local care pathways, and training physiotherapists to deliver it. Implementation theories and multifaceted implementation strategies will be used and adapted locally. The activities to evaluate the process include assessment of the implementation outcomes on healthcare professional and organizational levels, healthcare resource utilization and cost outcomes (1, 3 and 5 years) using registry data. In addition outcomes reported by patients participating in the GLA:D program will be collected at 3 months and 1, 3 and 10 years.

This project aims to bridge the gap between guideline-recommended OA-management and clinical practice. By implementing a systematic, evidence-based model of care, the study seeks to improve patient outcomes, reduce healthcare costs, and provide equitable access to care. The findings will inform future OA care strategies and will be disseminated and adapted to other healthcare contexts in Finland and can be adapted also internationally. The findings will be published in peer-reviewed journals and presented in national and international conferences.

ELIGIBILITY:
Data from national registries:

* Patients with diagnosed OA (ICD-10 / ICPC2)
* age over 18 years

Collection of GLA:D patient-reported outcomes:

Inclusion Criteria:

* Patients who are participating in theGLA:D program, diagnosed with hip or knee osteoarthritis, fluent in finnish
* age over 18 years

Exclusion Criteria:

* Other than OA-related cause of symptoms
* not able to answer the questionnaires in Finnish
* no access to a computer or mobile device to answer the questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: National registry data: Patients with diagnosed OA from all Wellbeing Services Counties in Finland
  GLA:D patient-reported outcome data: Patients who are participating in the GLA:D program, diagnosed with hip or knee osteoarthritis in any location that delivers GLA:D program.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Cost of OA care | 1 (primary endpoint), 3 and 5 years after implementation compared to baseline 2018-2024
  Healthcare cost associated with the new care pathway incluing annual healthcare consultation prevalence, number and cost of hospitalizations, OA-related surgical interventions and primary and specialized healthcare and outpatient specialist visits. Filled prescriptions, number and duration of OA-related sick leaves and disability pensions. Costs will be analysed using data from national registers in pre and post implementation, both within the pilot Wellbeing Services Counties and between the pilot and other Wellbeing Services Counties.
Reach: Proportion of patients directed according to the model of care | 1 (primary endpoint) 3 and 5 years after implementation
  Proportion of patients with hip and knee related symptoms and OA who contact healthcare that are referred to direct access physiotherapy and to GLA:D program

SECONDARY OUTCOMES:
Number of trained GLA:D trainers and physiotherapists | 1, 3 and 5 years after implementation
  Number of trained GLA:D trainers and physiotherapists in Finland, recorded in GLA:D Finland database by PI.
Participation of patients in GLA:D program | 1, 3 and 5 years after implementation
  Number of participants in GLA:D groups
Pain intensity during last week, numerical rating scale | Baseline, 3 months, 1, 3 and 10 years
  Numerical rating scale (NRS) 0-10, where 0 means no pain (better outcome) and 10 worst possible pain (worse outcome). a) worst pain b) average pain
Problems walking due to knee /hip | Baseline, 3 months, 1, 3 and 10 years
  yes / no
UCLA activity score | Baseline, 3 months, 1, 3 and 10 years
  UCLA activity score, 1= wholly inactive (worse outcome), 10 = regularly participate in impact sports (better outcome)
Fear of movement | Baseline, 3 months, 1, 3 and 10 years
  Are you afraid that your joints will be damaged from physical activity and exercise? yes / no
Use of painkillers | Baseline, 3 months, 1, 3 and 10 years
  Yes / no, and type of pain killers
Current employment | Baseline, 3 months, 1, 3 and 10 years
  Employed / student / unemployed / on sick leave full time / on sick leave part time / early retirement due to low ability to work / self-imposed early retirement / retired
Sick leave because of knee / hip during last year | Baseline, 3 months, 1, 3 and 10 years
  no / yes, under 1 month, yes 1-3 months, yes more than 3 months
EQ-5D-5L | Baseline, 3 months, 1, 3 and 10 years
  Mobility (1-5), self-care (1-5), usual activities (1-5), pain/ discomfort (1-5), anxiety / depression (1-5), eq-vas (0-100). Lower scores indicate a worse outcome.
K/HOOS-12 | Baseline, 3 months, 1, 3 and 10 years
  KOOS-12 asked if most affected joint is knee and HOOS-12 asked is most affected joint is hip. Scale 1-4 for each item, a lower score indicates a better outcome.
Global perceived effect | 3 months, 1, 3 and 10 years
  Much worse, an important worsening - much better an important improvement. 7-point likert scale, where a higher score indicates a better outcome.
Satisfaction with GLA:D | 3 and 12 months
  1-5 Not at all satisfied - very satisfied, higher score indicates a better outcome.
How often do you use what you've learned in GLA:D? | 3 months, 1, 3 and 10 years
  Never (1), every month (2), every week (3), every day (4), several times a day (5), a higher score indicates a better outcome.
Number of education and exercise sessions competed (face to face / online) | 3 months
  Numeral value
Falls over the last year | Baseline, 3 months, 1, 3 and 10 years
  Number of falls
Compliance in GLA:D program | 3 months
  Number of participated GLA:D sessions / participant.
Numbers of sites training / implementing GLA:D -program | 1, 3 and 5 years after implementation
  Number of sites training / implementing GLA:D -program in Finland. In numbers, based on documentation on GLA:D database by PI.
Number of GLA:D groups running | 1, 3 and 5 years after implementation
  Number of active GLA:D groups running, numbers, based on documentation on GLA:D Finland database by PI.
Modifications in the Model of care | 1, 3 and 5 years after implementation
  Descriptive qualitative reporting based on research diary: When and how modifactions in the Model of Care and Care pathways occured, whether it was unplanned or planned, reasons and goals for modification.

OTHER OUTCOMES:
The Determinants of Implementation Behaviour Questionnaire | after delivering first GLA:D program and at 12 months
  The multiprofessional version of Determinants of Implementation Behaviour Questionnaire (DIBQ-mp)
  Clinician reported determinants of implementation of guideline-based model of care and GLA:D program, designed according to the Theoretical Domains Framework. The items will be scored each separately on 7-point likert scale, where a lower score indicates that item being a barrier (worse outcome) and higher score towards facilitator (better outcome).
Gender | Baseline
  Male / female / other
Age | Baseline
  in years
Living situation | Baseline
  Living alone or with others
Educational level | Baseline
  Basic and vocational education
Medical comorbidities | Baseline
  High blood pressure and high cholesterol, Musculoskeletal conditions, Cardiovascular and blood diseases, Neurological diseases, Hormonal diseases, urinary diseasses, Gastrointestinal and liver diseases, Lung diseases, Cancer, Mental conditions, Diseases in the skin and other chronic diseases
Smoking | Baseline
  Smoking status
Duration of joint symptoms | Baseline
  Duration of joint symptoms in months / years
Most affected joint | Baseline, 1, 3 and 10 years
  Most affected joint (right/left hip, right/left knee)
Other affected joints | Baseline, 3 months, 1, 3 and 10 years
  Other affected joints (right/left hip, right/left knee)
Previous injury knee /hip | Baseline
  Previous injury that cuaused the person consult a doctor
Previous X-rays of affected joints | Baseline
  No / yes, more than 6 months ago / yes, within last 6 months / don't know
Osteoarthritis checklist | Baseline
  Knee: load related pain, reduced functional capacity, morning stiffness, crepitus, reduced knee movement, bony enlargement, age, sex, overweight, previous joint injury, occupational / recreational overuse / family members with osteoarthritis
  Hip: hip pain, stiffness after inactivity, reduced functional capacity, reduced hip flexion, reduced internal hip rotation, painful internal hip rotation, age, sex, overweight, previous joint injury, occupational / recreational overuse / family members with osteoarthritis
Previous and planned surgery of knee and hip | Baseline (previous and planned surgery), 3 months, 1, 3 and 10 years (planned surgery)
  Type and time of surgery
Short form of Orebro musculoskeletal pain screening questionnaire | Baseline, 3 months, 1, 3 and 10 years
  0-100 points, higher score indicates a higher risk (<40 points = low risk, 40-50 points = medium risk, >50 points = high risk)
Expectations on GLA:D program | Baseline
  1-5 1= very large / complete improvement, 5 = Very small or no improvement

IPD SHARING:
Plan to Share IPD: No